CLINICAL TRIAL: NCT03194971
Title: NovoTTF Treatment Signatures in Glioblastoma Patients At Autopsy
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Peter LaViolette, Principal Investigator, Medical College of Wisconsin
Other Study IDs: PRO00017446
Record Dates: First submitted 2017-06-12; First posted 2017-06-21 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
Keywords: glioblastoma; brain tumor autopsy; autopsy; Optune therapy; tumor treatment fields; TTFields; Recurrent glioblastoma; grade IV; brain tumor; newly diagnosed glioblastoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Samples are obtained from regions suspicious for tumor at autopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TTField at Recurrence
  Interventions: Device: Tumor samples from patients treated with TTFields at tumor recurrence.
- TTField at New Diagnosis
  Interventions: Other: Tumor samples from patients treated with TTFields at initial diagnosis.

INTERVENTIONS:
Other: Tumor samples from patients treated with TTFields at initial diagnosis. — Pathological assessment of tumor cellularity, apoptosis, and quantitative histo-morphometry of residual tumor cells will be performed. Each metric will be statistically compared between groups.
  Groups: TTField at New Diagnosis
Device: Tumor samples from patients treated with TTFields at tumor recurrence. — Pathological assessment of tumor cellularity, apoptosis, and quantitative histo-morphometry of residual tumor cells will be performed. Each metric will be statistically compared between groups.
  Groups: TTField at Recurrence

SUMMARY:
This study will assess whole brain samples from glioblastoma patients at autopsy to determine the underlying pathological signatures of tumor treatment fields at autopsy.

DETAILED DESCRIPTION:
RATIONALE:

Optune therapy with tumor treatment fields (TTFields) has recently been FDA approved for the treatment of newly diagnosed glioblastoma due to a recent clinical trial that showed improvement in progression free survival and overall survival compared to standard therapy. (1) TTFields also have a role in the recurrent glioblastoma treatment where it has demonstrated equal efficacy to second-line chemotherapy also has been shown to tumor progression and improve overall survival.(2) Though preclinical studies are ongoing, glioblastoma patients who have undergone TTField therapy have not yet been assessed at autopsy to determine both the pathological signature of TTField treatment, and the pattern of failure. This study will determine how the underlying pathological signatures of tumors treated with TTFields differ from those naïve to TTFields by comparing tumor tissue at autopsy.

STUDY:

All patients undergoing TTField therapy for newly diagnosed and recurrent glioblastoma will be considered for inclusion for this study. The investigators expect to enroll five patients per year for four years, totaling 10 patients treated upfront and 10 patients treated at tumor recurrence. An objective of this study is to determine differences in the pathological pattern of failure when patients are treated with TTFields at initial diagnosis (up-front) compared to those treated at tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma, World Health Organization (WHO) grade IV, patients undergoing TTField therapy.
* Recurrent glioblastoma WHO grade IV, patients undergoing TTField therapy.

Exclusion Criteria:

* TTField compliance < 75%.
* Any contraindication to Optune TTField treatment.
* Initial brain tumor diagnosis < WHO grade IV.
* Duration of TTField therapy < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly Diagnosed Glioblastoma Patients undergoing standard of care treatment consisting of surgery followed by chemo-radiation therapy will have the addition of Optune TTField therapy together with adjuvant chemotherapy. OR Recurrent Glioblastoma Patients with glioblastoma tumor recurrence defined by either imaging criteria, or deteriorating neurological function will be offered Optune TTField treatment at the discretion of the neurooncologist.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of mitotically active cells | At baseline
  Tissue samples will be obtained at autopsy and stained for KI-67. Slides will then be digitized, and the number of active cells will be counted computationally.
Number of mitotically inactive cells | At baseline
  Tissue samples will be obtained at autopsy and stained for KI-67. Slides will then be digitized, and the number of not active cells will be counted computationally.
Mitotic Ratio | At baseline
  Number of mitotically active cells divided by the number of not mitotically active cells per patient will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Peter LaViolette, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No